CLINICAL TRIAL: NCT03978832
Title: An Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of 180 mg Risperidone Subcutaneous Injection (PERSERIS) Following a Switch From 6 mg Oral Risperidone in Patients With Clinically Stable Schizophrenia
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of 180 mg Subcutaneous Risperidone From 6 mg Oral Risperidone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDV-7000-401
Record Dates: First submitted 2019-05-30; First posted 2019-06-07 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Intervention Model Description: The study will enroll subjects currently on a stable dose of 5 or 6 mg of oral risperidone. After screening, eligible subjects will be admitted to the clinical unit and stabilized on 6 mg daily (3 mg oral risperidone twice a day) for 5 days, followed by an additional 3 days, during which the first injection of PERSERIS will be administered. Subjects will then return to the clinical unit every 28 days for an additional 3 admit periods for subsequent PERSERIS injections (2 injections per visit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Risperidone followed by PERSERIS (Experimental): All subjects will receive 2 SC injections of PERSERIS at each study visit every 28 days for a total of 4 visits of 2 injections each. The first 3 visit injections will be administered in the abdomen and the final visit injections will be administered in the back of the upper arm.
  Interventions: Drug: PERSERIS; Drug: Risperidone

INTERVENTIONS:
Drug: PERSERIS — PERSERIS is an extended-release SC injectable suspension administered once-monthly
  Other Names: long acting risperidone
Drug: Risperidone — Oral risperidone
  Other Names: Risperdal

SUMMARY:
This study evaluates PERSERIS at a higher dose than what has been administered in previous clinical trials. Subjects with stable schizophrenia on a dose of 5-6 mg oral risperidone will be switched to PERSERIS at the higher dose, which is believed to be similar to the oral dose

DETAILED DESCRIPTION:
PERSERIS is an extended-release subcutaneous (SC) injectable suspension administered monthly for the treatment of schizophrenia in adults. PERSERIS was approved by the FDA at doses equivalent to 3 mg and 4 mg oral risperidone. Many patients require doses of 5-6 mg oral risperidone and above, and this study will test a higher dose of PERSERIS in order to meet this need.

Eligible subjects will initially be stabilized in the clinical unit on 6 mg oral risperidone for 5 days and transition to an approximate dose of PERSERIS by SC injection. PERSERIS will be administered every 28 days and subjects will be admitted to the clinical unit the day before, and remain in the unit for 3 days after each injection for pharmacokinetics (PK) and safety evaluations (a total of 8 days for the first injection including the stabilization period). Subjects will return to the clinic between injections for additional PK, safety and efficacy assessments at scheduled intervals until the next injection.

A total of 4 doses of PERSERIS will be administered. The 4th dose will evaluate an alternate site for injection, and will be administered in the back of the upper arm.

Subjects will return to the clinical unit for an end of study visit and will receive a follow up phone call to assess for adverse events one week after the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Clinically stable as defined as no hospitalizations for acute exacerbations within 3 months of screening and Screening PANSS score ≤70
* Total body mass index (BMI) between 18 and 35 kg/m2
* Given written informed consent

Exclusion Criteria:

* Received a once-monthly long-acting injectable (LAI) antipsychotic within 60 days of screening and a once every 3 month LAI antipsychotic within 120 days of screening
* Taking the following concurrent or over the counter (OTC) products:

  1. Inducers or inhibitors of CYP2D6 within 14 days or 5 half-lives whichever is greater prior to study screening
  2. Bupropion, chlorpheniramine, cimetidine, clomipramine, doxepin or quinidine within 30 days prior to study screening
  3. Clozapine, phenothiazines, aripiprazole, haloperidol or any other antipsychotic other than oral risperidone within 14 days prior to study screening
  4. Selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRIs) within 30 days prior to study screening
  5. Opioids or opioid-containing analgesics within 14 days prior to study screening
  6. Medications, in the addition to those listed above which in the opinion of the Investigator in conjunction with the medical monitor, may be expected to significantly interfere with the metabolism or excretion of risperidone and/or 9-hydroxyrisperidone, that may be associated with a significant drug interaction with risperidone, or that may pose a significant risk to subjects' participation in the study. The medical monitor should be contacted with any questions regarding the use of CYP2D6 or 3A4 inducers or inhibitors in particular.
* History of cancer (with the exception of resected basal cell or squamous cell carcinoma of the skin) unless they have been disease free for ≥5 years.
* Another active medical condition or organ disease that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug.
* Evidence or history of a significant hepatic disorder that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug. Individuals with acute or chronic hepatitis (including but not limited to hepatitis B or C); or individuals with 1) total bilirubin >1.5x the upper limit of normal (ULN) and/or 2) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3x ULN will be excluded.
* A history of renal disease, or a creatinine clearance of less than 60 mL/min (as determined by the Cockcroft-Gault formula).
* A history of orthostatic hypotension, syncope, significant low white blood cell (WBC) count (i.e., based on absolute neutrophil count or drug-induced leukopenia or other medical conditions including, but not limited to, history of heart attack (i.e., myocardial infarction) or brain injury (i.e., traumatic with loss of consciousness and/or cardiovascular accident) within a year of Screening and clinically significant low blood pressure or arrhythmias as interpreted by the principal investigator (PI).
* Corrected QT interval [Fridericia's calculation (QTcF)] >450 msec (male) or >470 msec (female) at screening or prior to administration of the 1st dose of PERSERIS, or with a known history of Torsades de Points, or family member with sudden unexplained cardiac death.
* Known to have AIDS (acquired immunodeficiency syndrome) or to be HIV (human immunodeficiency virus) positive.
* Suicidal ideation with intent and plan, as assessed by affirmative answers to C-SSRS questions 4 and 5 of the ideation section,or suicide attempts within the last 6 months as noted on the C-SSRS, or subjects with uncontrolled depression in the opinion of the Investigator.
* Known diagnosis of type 1 diabetes or subjects with Haemoglobin A1c (HbA1c) >8.0% at screening.
* Participated in a clinical trial within 30 days prior to study screening.
* Significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.
* Meet the criteria for the diagnosis of current moderate or severe substance use disorder.
* Prior allergic reactions, sensitivities, or other known contraindications to any component of PERSERIS.
* Women of childbearing potential who are pregnant or breastfeeding, seeking pregnancy or failing to use adequate contraceptive methods during the study.
* Positive urine drug screen (UDS) anytime through Day -1 for opioids, cocaine, amphetamines, methadone, cannabinoids, barbiturates, benzodiazepines, methamphetamine and phencyclidine, unless the positive screen is determined to be secondary to an allowable concomitant medication. If a positive UDS is possibly the result of a subject's use of OTC or prescription medications, a repeat urine drug screen may be permissible. Study site personnel should contact the medical monitor for approval to retest.
* Tardive dyskinesia as assessed by a score of ≥2 on Item 8 of the Abnormal Involuntary Movement Scale (AIMS) at Screening.
* Epilepsy or other seizure disorders, Parkinson's disease or dementia.
* History of neuroleptic malignant syndrome.
* Previously injected with PERSERIS within 6 months prior to screening.
* Unable, in the opinion of the PI, to comply fully with the study requirements.
* Determined to be poor metabolisers, intermediate metabolisers or ultra-rapid metabolisers for CYP2D6 genotype.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, Principal Investigator — Collaborative Neuroscience Network
Locations (1):
- Collaborative Neuroscience Network, Garden Grove, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walling DP, Shinde SN, Pogoda JM, Kharidia J, Laffont CM. An Open-Label Study to Assess Monthly Risperidone Injections (180 mg) Following Switch from Daily Oral Risperidone (6 mg) in Stable Schizophrenic Patients. Clin Drug Investig. 2024 Apr;44(4):251-260. doi: 10.1007/s40261-024-01347-1. Epub 2024 Feb 22. PMID 38388986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants from the community between June and December 2019. Participants were on a stable dose of 5 mg or 6 mg of oral risperidone daily; any daily or twice daily dosing combination was acceptable.
Pre-assignment Details: After providing informed consent potential participants were screened, and after eligibility was confirmed, participants were stabilized on 6 mg daily of oral risperidone (3 mg administered twice a day [BID] approximately 12 hours apart) for 5 days.
  After completion of the stabilization period, participants were eligible to receive 180 mg PERSERIS (subcutaneous risperidone), administered as two 90 mg SC injections every 28 days.
Groups:
- Oral Risperidone Followed by PERSERIS: All participants received up to 4 monthly doses of 180 mg PERSERIS (each 180 mg dose was administered as two 90 mg SC injections). The first 3 monthly doses were administered in the abdominal region while the fourth monthly dose was administered in the back of the upper arm.
  PERSERIS: PERSERIS (subcutaneous risperidone) is an extended-release SC injectable suspension administered once-monthly
  Risperidone: Oral risperidone
Period: Overall Study
Arm/Group | Oral Risperidone Followed by PERSERIS
Started | 69 (69 participants signed the ICF and entered screening; 25 met eligibility criteria and were enrolled.)
Stabilization Period | 25
Treatment Period | 23
Completed | 15
Not Completed | 54
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2
Not completed — did not pass screening criteria | 44

BASELINE CHARACTERISTICS:
Population: The baseline number is the number of participants who received oral risperidone during the stabilization period and at least one PERSERIS injection. This equals the number of participants included in the safety and efficacy populations. There was one additional participant included in the PK population who had PK data from oral risperidone but did not receive PERSERIS and was not included in the safety population.
Groups:
- Oral Risperidone Followed by PERSERIS: All participants received up to 4 monthly doses of 180 mg PERSERIS (each 180 mg dose was administered as two 90 mg SC injections). The first 3 monthly doses were administered in the abdominal region while the fourth monthly dose was administered in the back of the upper arm.
  PERSERIS: PERSERIS is an extended-release SC injectable suspension administered once-monthly
  Risperidone: Oral risperidone
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.49 (4.650)
CYP2D6 Genotype [Count of Participants; unit: Participants] — CYP2D6 was analyzed for the purpose of assessing genetic variation in enzymes that may affect the concentration of PERSERIS, and therefore its safety and efficacy. Depending on the result of the analysis, patients were classified as ultrarapid, extensive, intermediate or poor metabolizers of CYP2D6, with extensive metabolizers being considered as normal metabolism. Altered metabolism of CYP2D6 may lead to concentrations of risperidone (the active ingredient in PERSERIS) outside the recommended therapeutic range, increasing the risk of treatment failure or side effects.
  Participants
    Poor | 0
    Intermediate | 0
    Extensive | 23
    Ultra-rapid | 0

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Average Plasma Concentration (Cavg,ss) of Risperidone and Total Active Moiety
Description: Cavg,ss for risperidone and total active moiety after oral and SC administration
Time Frame: 0-12 hours post-dose on Day -1, and 0-672 hours after Dose 3
Population: The primary PK analysis was conducted in participants who received at least 3 doses of PERSERIS 180 mg and provided adequate blood samples for the determination of Cavg after the third dose (primary PK population).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 16
ng/mL
  Risperidone after oral dosing | 5.150 (43.3)
  Risperidone after Dose 3 | 10.200 (65.3)
  Total active moiety after oral dosing | 43.730 (34.8)
  Total active moiety after Dose 3 | 44.049 (24.4)

2. Secondary Outcome: Assessment of Local Injection Site Tolerability*
Description: Injection site tolerability was measured by injection site grading for redness, induration, swelling and tenderness/pain. These were graded on a scale from 0 to 4 for severity (none, mild, moderate, severe and potentially life-threatening)
Time Frame: First injection at Day 1 until last injection administered at Day 85
Population: The number of participants assessed is the actual number who received the injection at each visit. *By the nature of this outcome measure (injection site), all results are reported for participants who had received PERSERIS
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants
  Dose 1 injection site pain grade: None | 22
  Dose 1 injection site pain grade: Mild | 1
  Dose 2 injection site pain grade: number analyzed (Participants) | 20
  Dose 2 injection site pain grade: None | 19
  Dose 2 injection site pain grade: Mild | 1
  Dose 3 injection site pain grade: number analyzed (Participants) | 16
  Dose 3 injection site pain grade: None | 16
  Dose 3 injection site pain grade: Mild | 0
  Dose 4 injection site pain grade: number analyzed (Participants) | 16
  Dose 4 injection site pain grade: None | 15
  Dose 4 injection site pain grade: Mild | 1
  Dose 1 injection site tenderness grade: None | 21
  Dose 1 injection site tenderness grade: Mild | 2
  Dose 2 injection site tenderness grade: number analyzed (Participants) | 20
  Dose 2 injection site tenderness grade: None | 18
  Dose 2 injection site tenderness grade: Mild | 2
  Dose 3 injection site tenderness grade: number analyzed (Participants) | 16
  Dose 3 injection site tenderness grade: None | 15
  Dose 3 injection site tenderness grade: Mild | 1
  Dose 4 injection site tenderness grade: number analyzed (Participants) | 16
  Dose 4 injection site tenderness grade: None | 13
  Dose 4 injection site tenderness grade: Mild | 3
  Dose 1 injection site erythema/redness grade: None | 22
  Dose 1 injection site erythema/redness grade: Mild | 1
  Dose 2 injection site erythema/redness grade: number analyzed (Participants) | 20
  Dose 2 injection site erythema/redness grade: None | 20
  Dose 2 injection site erythema/redness grade: Mild | 0
  Dose 3 injection site erythema/redness grade: number analyzed (Participants) | 16
  Dose 3 injection site erythema/redness grade: None | 16
  Dose 3 injection site erythema/redness grade: Mild | 0
  Dose 4 injection site erythema/redness grade: number analyzed (Participants) | 16
  Dose 4 injection site erythema/redness grade: None | 16
  Dose 4 injection site erythema/redness grade: Mild | 0
  Dose 1 injection site induration/swelling grade: None | 23
  Dose 1 injection site induration/swelling grade: Mild | 0
  Dose 2 injection site induration/swelling grade: number analyzed (Participants) | 20
  Dose 2 injection site induration/swelling grade: None | 20
  Dose 2 injection site induration/swelling grade: Mild | 0
  Dose 3 injection site induration/swelling grade: number analyzed (Participants) | 16
  Dose 3 injection site induration/swelling grade: None | 15
  Dose 3 injection site induration/swelling grade: Mild | 1
  Dose 4 injection site induration/swelling grade: number analyzed (Participants) | 16
  Dose 4 injection site induration/swelling grade: None | 14
  Dose 4 injection site induration/swelling grade: Mild | 2

3. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Local Injection Site*
Description: The injection site was evaluated for adverse events by observation and examination by appropriately trained personnel.
Time Frame: First injection at Day 1 until Day 120
Population: *By the nature of this outcome measure (injection site), all results are reported for participants who had received PERSERIS
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants | 1

4. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Changes in Vital Signs
Description: Vital sign measurement was performed, including orthostatic blood pressure, and clinically significant changes were reported as adverse events (AE). Vital sign measurement also included measurement of pulse rate, oral temperature and respiratory rate. Determination of whether the changes were AEs was made by the investigator or a medically qualified designee. If determined to be an AE, the measurement was repeated at appropriate intervals until the value returned to an acceptable range and the subject was clinically stable, a specific diagnosis was established, or the condition otherwise explained.
Time Frame: Time subjects sign the informed consent form throughout the study until EOS (Day 113)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants | 1

5. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Changes in ECG
Description: ECGs were performed, and clinically significant changes in parameters were reported as adverse events (AE). ECGs were performed after 5 minutes of rest, and ECG parameters including QT interval, PR interval, QRS interval and heart rate was recorded. The ECG measurements were evaluated during the visit and determination of whether any abnormalities were AEs was made by the investigator or a medically qualified designee. If determined to be an AE, the measurement was repeated at appropriate intervals until the value returned to an acceptable range and the subject was clinically stable, a specific diagnosis was established, or the condition otherwise explained.
Time Frame: Time participants sign the informed consent form throughout the study until EOS (Day 113)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants | 0

6. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Changes in Body Weight
Description: Body weight, with shoes off, was measured and clinically significant changes in weight was reported as adverse events (AE). Determination of whether the changes were AEs was made by the investigator or a medically qualified designee. If determined to be an AE, the measurement was repeated at appropriate intervals until the value returned to an acceptable range and the subject was clinically stable, a specific diagnosis was established, or the condition otherwise explained.
Time Frame: Time subjects sign the informed consent form throughout the study until EOS (Day 113)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants | 1

7. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Changes in Laboratory Testing
Description: Laboratory testing was performed by the local clinical laboratory accredited by the College of American Pathologists, and clinically significant changes from baseline were reported as AEs. Subjects were expected to fast for a minimum of 8 hours prior to blood draws for all laboratory assessments except at the screening visit. Prior to entering the study, any abnormal laboratory test results were to be considered not clinically significant. Any abnormal hematology, serum chemistry or urinalysis test result after study drug intake that was determined by the investigator or a medically qualified designee to be clinically significant was reported as an AE. If determined to be an AE, the measurement was repeated at appropriate intervals until the value returned to an acceptable range or it was determined that resolution was not expected.
Time Frame: Time subjects sign the informed consent form throughout the study until end of study (EOS) visit (Day 113)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants | 3

8. Secondary Outcome: The Number of Participants With TEAEs as Assessed by Extrapyramidal Symptoms (EPS) of Anti-psychotic Drug Treatment
Description: Safety of treatment was measured by administration of symptom questionnaires including AIMS, Barnes Akathisia Rating Scale (BARS) and Simpson-Angus Scale (SAS), as well as by assessment by the investigator or suitably qualified medical designee. The AIMS is a tool that aids in early detection and ongoing monitoring of tardive dyskinesia, a movement disorder. The BARS is a 4-item scale that detects the presence and severity of any drug-induced restlessness. The SAS is a 10-item scale used to detect the presence of drug-induced Parkinsonism (movement disorder seen in Parkinson's disease) and extrapyramidal side effects and evaluates symptom severity. Extrapyramidal symptoms include involuntary or uncontrollable movements, tremors, and muscle contractions.
Time Frame: Time subjects sign the informed consent form throughout the study until EOS (Day 113)
Population: There were no clinically important differences in mean scores across study visits. TEAEs related to EPS are reported below
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants
  Akathisia | 1
  Dyskinesia | 2
  Parkinsonian gait | 1
  Tremor | 1

9. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: Clinical outcome (efficacy endpoint) as measured by change from baseline in PANSS scores was measured. PANSS is a medical scale designed to measure schizophrenia symptom severity utilizing a 30 item, 7-point rating scheme. The PANSS Is scored by a summation of ratings across items, with a total potential range of 7-210; higher results indicate greater severity of illness.
  Only total score changes from baseline are reported here.
Time Frame: Baseline, defined as last assessment prior to first injection, through Day 113 (EOS)
Population: PANSS total scores change from baseline measure from baseline through Day 113 for those participants with results reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
score on a scale
  Total score change from baseline: Dose 1 Day 2 | -0.2 (3.52)
  Total score change from baseline: Dose 1 Day 8 | 0.9 (3.91)
  Total score change from baseline: Dose 1 Day 15: number analyzed (Participants) | 22
  Total score change from baseline: Dose 1 Day 15 | 0.7 (4.81)
  Total score change from baseline: Dose 1 Day 22: number analyzed (Participants) | 22
  Total score change from baseline: Dose 1 Day 22 | -0.4 (4.16)
  Total score change from baseline: Dose 2 Day 29: number analyzed (Participants) | 22
  Total score change from baseline: Dose 2 Day 29 | -0.9 (5.05)
  Total score change from baseline: Dose 2 Day 50: number analyzed (Participants) | 19
  Total score change from baseline: Dose 2 Day 50 | -0.5 (7.21)
  Total score change from baseline: Dose 3 Day 57: number analyzed (Participants) | 16
  Total score change from baseline: Dose 3 Day 57 | -2.9 (4.92)
  Total score change from baseline: Dose 4 Day 85: number analyzed (Participants) | 16
  Total score change from baseline: Dose 4 Day 85 | -0.9 (6.00)
  Total score change from baseline: Day 113-EOS: number analyzed (Participants) | 14
  Total score change from baseline: Day 113-EOS | 1.6 (6.22)

10. Secondary Outcome: Clinical Global Impression-Severity of Illness Scale (CGI-S)
Description: Clinical outcome (efficacy endpoint) as measured by change from baseline in CGI-S scores was measured. The CGI-S is a measurement of the total severity of illness where one question is assessed. Responses range from 0 (not assessed) to 7 (most extremely ill).
Time Frame: Baseline through EOS (Day 113)
Population: Severity of illness observed values were measured and change from baseline calculated for those participants with results reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
score on a scale
  Change from baseline: Dose 1/Day 2 | -0.1 (0.29)
  Change from baseline: Dose 1/Day 8 | 0.0 (0.21)
  Change from baseline: Dose 1/Day 15: number analyzed (Participants) | 22
  Change from baseline: Dose 1/Day 15 | 0.0 (0.38)
  Change from baseline: Dose 1/Day 22: number analyzed (Participants) | 22
  Change from baseline: Dose 1/Day 22 | 0.0 (0.44)
  Change from baseline: Dose 2/Day 29: number analyzed (Participants) | 22
  Change from baseline: Dose 2/Day 29 | 0.0 (0.44)
  Change from baseline: Dose 2/Day 50: number analyzed (Participants) | 19
  Change from baseline: Dose 2/Day 50 | 0.0 (0.47)
  Change from baseline: Dose 3/Day 57: number analyzed (Participants) | 16
  Change from baseline: Dose 3/Day 57 | 0.1 (0.44)
  Change from baseline: Dose 4/Day 85: number analyzed (Participants) | 16
  Change from baseline: Dose 4/Day 85 | 0.1 (0.50)
  Change from baseline: EOS/Day 113: number analyzed (Participants) | 14
  Change from baseline: EOS/Day 113 | 0.0 (0.55)

11. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)-Change
Description: Significant changes from baseline in C-SSRS scores were reported as adverse events. The C-SSRS is based on a categorization of thoughts and behavior that are identified as related to suicidal behavior. The scale captures the occurrence, severity and frequency of suicide related thoughts and behaviors throughout lifetime at screening and for the time interval since last administration during a study. Responses are indicated as yes (thought or behavior did occur) or no (thought or behavior did not occur). If a yes response is received, then follow up questions are asked. The outcome of the C-SSRS is a numerical score obtained from each of the categories. Scores can range from 0-25, indicating the intensity rating, and any score greater than 0 may indicate the need for mental health intervention. Higher scores indicate greater intensity (i.e. worse outcome).
Time Frame: Screening through EOS (Day 113)
Population: Only actual number of participants assessed at visit was reported. Only change in suicidal behavior from baseline at Dose 1/Day 8 (first measure after baseline) and EOS is reported as all numbers are zero.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
score on a scale
  Change in Maximum Suicidal Ideation at Dose 1/Day 8 | 0.0 (0.00)
  Change in Maximum Suicidal Ideation at EOS: number analyzed (Participants) | 14
  Change in Maximum Suicidal Ideation at EOS | 0.0 (0.00)
  Change in Suicidal Ideation Intensity Score at Dose 1/Day 8 | 0.0 (0.00)
  Change in Suicidal Ideation Intensity Score at EOS: number analyzed (Participants) | 14
  Change in Suicidal Ideation Intensity Score at EOS | 0.0 (0.00)
  Change in Maximum Suicidal Behavior at Dose 1/Day 8: number analyzed (Participants) | 22
  Change in Maximum Suicidal Behavior at Dose 1/Day 8 | 0.0 (0.00)
  Change in Maximum Suicidal Behavior at EOS: number analyzed (Participants) | 14
  Change in Maximum Suicidal Behavior at EOS | 0.0 (0.00)

12. Secondary Outcome: Safety as Measured by Columbia-Suicide Severity Rating Scale (C-SSRS) Scores
Description: Safety of treatment was measured by characterization of thoughts and behavior related to suicidal behavior. This was assessed by administration of the C-SSRS at designated visits. The scale captures the occurrence, severity and frequency of suicide related thoughts and behaviours throughout lifetime at screening and for the time interval since last administration during a study. Questions solicit the type of information needed to determine if a suicide-related thought or behavior occurred.
Time Frame: Screening through EOS (Day 113)
Population: Only actual number of participants assessed at visit was reported. Only results for lifetime, past 6 months and EOS are reported as all responses are 'no' after lifetime.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 23
Participants
  Any Suicidal Ideation - Lifetime: No | 15
  Any Suicidal Ideation - Lifetime: Yes | 8
  Any Suicidal Ideation - Past 6 months: No | 23
  Any Suicidal Ideation - Past 6 months: Yes | 0
  Any Suicidal Ideation - EOS: number analyzed (Participants) | 14
  Any Suicidal Ideation - EOS: No | 14
  Any Suicidal Ideation - EOS: Yes | 0
  Any Suicidal Behavior - Lifetime: No | 17
  Any Suicidal Behavior - Lifetime: Yes | 6
  Any Suicidal Behavior - Past 6 months: number analyzed (Participants) | 20
  Any Suicidal Behavior - Past 6 months: No | 20
  Any Suicidal Behavior - Past 6 months: Yes | 0
  Any Suicidal Behavior - EOS: number analyzed (Participants) | 14
  Any Suicidal Behavior - EOS: No | 14
  Any Suicidal Behavior - EOS: Yes | 0
  Any Suicidal Ideation or Behavior - Lifetime: No | 15
  Any Suicidal Ideation or Behavior - Lifetime: Yes | 8
  Any Suicidal Ideation or Behavior - Past 6 months: number analyzed (Participants) | 20
  Any Suicidal Ideation or Behavior - Past 6 months: No | 20
  Any Suicidal Ideation or Behavior - Past 6 months: Yes | 0
  Any Suicidal Ideation or Behavior - EOS: number analyzed (Participants) | 14
  Any Suicidal Ideation or Behavior - EOS: No | 14
  Any Suicidal Ideation or Behavior - EOS: Yes | 0

13. Secondary Outcome: Minimum Plasma Concentration Over the Dosing Interval
Description: Minimum observed plasma concentration of risperidone, 9-hydroxyrisperidone (9-OH) and total active moiety over the dosing interval after oral dosing and SC doses 1, 3 and 4
Time Frame: Calculated over the dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4).
Population: PK population. Actual number of participants analyzed for each period is reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
ng/mL
  Risperidone after oral dosing | 1.066 (89.0)
  Risperidone after Dose 1: number analyzed (Participants) | 20
  Risperidone after Dose 1 | 3.017 (39.0)
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 4.519 (48.1)
  Risperidone after Dose 4: number analyzed (Participants) | 14
  Risperidone after Dose 4 | 5.020 (48.7)
  9-OH after oral dosing | 27.705 (41.7)
  9-OH after Dose 1: number analyzed (Participants) | 20
  9-OH after Dose 1 | 13.922 (63.6)
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 16.951 (41.6)
  9-OH after Dose 4: number analyzed (Participants) | 14
  9-OH after Dose 4 | 14.820 (46.3)
  Total active moiety after oral dosing | 28.329 (39.6)
  Total active moiety after Dose 1: number analyzed (Participants) | 20
  Total active moiety after Dose 1 | 17.852 (55.8)
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 22.250 (37.7)
  Total active moiety after Dose 4: number analyzed (Participants) | 14
  Total active moiety after Dose 4 | 22.063 (35.7)

14. Secondary Outcome: Maximum Plasma Concentration Over the Dosing Interval
Description: Maximum observed plasma concentration of risperidone, 9-hydroxyrisperidone (9-OH) and total active moiety over the dosing interval after oral dosing and SC doses 1, 3 and 4
Time Frame: Calculated over the dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4)
Population: Analysis population is the PK population. Actual number of participants analyzed for each period is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
ng/mL
  Risperidone after oral dosing | 14.052 (45.2)
  Risperidone after Dose 1: number analyzed (Participants) | 22
  Risperidone after Dose 1 | 16.743 (57.1)
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 18.635 (54.6)
  Risperidone after Dose 4: number analyzed (Participants) | 15
  Risperidone after Dose 4 | 29.821 (65.1)
  9-OH after oral dosing | 45.464 (40.0)
  9-OH after Dose 1: number analyzed (Participants) | 22
  9-OH after Dose 1 | 45.285 (43.3)
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 56.476 (34.5)
  9-OH after Dose 4: number analyzed (Participants) | 15
  9-OH after Dose 4 | 52.240 (27.4)
  Total active moiety after oral dosing | 58.453 (33.5)
  Total active moiety after Dose 1: number analyzed (Participants) | 22
  Total active moiety after Dose 1 | 58.317 (38.4)
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 70.597 (30.7)
  Total active moiety after Dose 4: number analyzed (Participants) | 15
  Total active moiety after Dose 4 | 77.219 (32.5)

15. Secondary Outcome: Percent Fluctuation in Concentration Over the Dosing Interval
Description: Plasma concentration variation of risperidone, 9-OH and total active moiety over the dosing interval was measured by percent fluctuation after oral dosing and SC doses 1, 3 and 4 at steady state.
Time Frame: Calculated over the dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4)
Population: PK population. Actual number of participants analyzed for each period is reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of fluctuation
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
percentage of fluctuation
  Risperidone after oral dosing | 253.335 (33.6)
  Risperidone after Dose 1: number analyzed (Participants) | 20
  Risperidone after Dose 1 | 174.653 (35.4)
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 135.267 (19.6)
  Risperidone after Dose 4: number analyzed (Participants) | 14
  Risperidone after Dose 4 | 190.117 (66.7)
  9-OH after oral dosing | 46.787 (32.0)
  9-OH after Dose 1: number analyzed (Participants) | 20
  9-OH after Dose 1 | 115.645 (48.1)
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 115.286 (55.5)
  9-OH after Dose 4: number analyzed (Participants) | 14
  9-OH after Dose 4 | 116.852 (44.7)
  Total active moiety after oral dosing | 71.468 (26.0)
  Total active moiety after Dose 1: number analyzed (Participants) | 20
  Total active moiety after Dose 1 | 115.113 (29.2)
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 106.210 (28.6)
  Total active moiety after Dose 4: number analyzed (Participants) | 14
  Total active moiety after Dose 4 | 118.435 (34.5)

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval
Description: Area under the plasma concentration-time curve (AUC) was measured for risperidone, 9-OH and total active moiety.
Time Frame: Calculated over the dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4).
Population: PK population; actual number of participants analyzed for each period is reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
hr*ng/mL
  Risperidone after oral dosing | 60.354 (54.4)
  Risperidone after Dose 1: number analyzed (Participants) | 20
  Risperidone after Dose 1 | 5021.191 (55.0)
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 6854.855 (65.2)
  Risperidone after Dose 4: number analyzed (Participants) | 14
  Risperidone after Dose 4 | 7762.268 (63.6)
  9-OH after oral dosing | 432.801 (38.4)
  9-OH after Dose 1: number analyzed (Participants) | 20
  9-OH after Dose 1 | 17615.97 (44.0)
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 22203.31 (28.9)
  9-OH after Dose 4: number analyzed (Participants) | 14
  9-OH after Dose 4 | 20527.19 (30.2)
  Total active moiety after oral dosing | 489.888 (34.0)
  Total active moiety after Dose 1: number analyzed (Participants) | 20
  Total active moiety after Dose 1 | 22955.74 (37.5)
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 29602.72 (24.4)
  Total active moiety after Dose 4: number analyzed (Participants) | 14
  Total active moiety after Dose 4 | 29217.83 (23.4)

17. Secondary Outcome: Average Plasma Concentration (Cavg) Over the Dosing Interval of Risperidone, 9-OH and Total Active Moiety
Description: Average plasma concentration of risperidone, 9-hydroxyrisperidone (9-OH) and total active moiety over the dosing interval after oral dosing and SC doses 1, 3 and 4.
Time Frame: Calculated over the dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4).
Population: PK population; actual number of participants analyzed for each period is reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
ng/mL
  Risperidone after oral dosing | 5.030 (54.4)
  Risperidone after Dose 1: number analyzed (Participants) | 20
  Risperidone after Dose 1 | 7.454 (55.2)
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 10.200 (65.3)
  Risperidone after Dose 4: number analyzed (Participants) | 14
  Risperidone after Dose 4 | 11.618 (63.2)
  9-OH after oral dosing | 36.066 (38.4)
  9-OH after Dose 1: number analyzed (Participants) | 20
  9-OH after Dose 1 | 26.148 (44.0)
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 33.039 (28.8)
  9-OH after Dose 4: number analyzed (Participants) | 14
  9-OH after Dose 4 | 30.723 (31.3)
  Total active moiety after oral dosing | 40.823 (34.0)
  Total active moiety after Dose 1: number analyzed (Participants) | 20
  Total active moiety after Dose 1 | 34.077 (37.5)
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 44.049 (24.4)
  Total active moiety after Dose 4: number analyzed (Participants) | 14
  Total active moiety after Dose 4 | 43.729 (24.0)

18. Secondary Outcome: Trough Plasma Concentration
Description: Trough (pre-dose) plasma concentrations were measured for risperidone, 9-OH and total active moiety for SC doses 1, 3 and 4
Time Frame: Calculated over the dosing interval (0-672 hours) after Dose 1, 3 or 4.
Population: PK population; actual number of participants analyzed for each period is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
ng/mL
  Risperidone after Dose 1 | 1.766 (117.9)
  Risperidone after dose 3: number analyzed (Participants) | 16
  Risperidone after dose 3 | 5.066 (48.0)
  Risperidone after Dose 4: number analyzed (Participants) | 16
  Risperidone after Dose 4 | 4.966 (62.9)
  9-OH after dose 1 | 33.696 (37.9)
  9-OH after dose 3: number analyzed (Participants) | 16
  9-OH after dose 3 | 20.326 (51.0)
  9-OH after dose 4: number analyzed (Participants) | 16
  9-OH after dose 4 | 17.983 (39.2)
  Total active moiety after dose 1: number analyzed (Participants) | 23
  Total active moiety after dose 1 | 35.553 (35.6)
  Total active moiety after dose 3: number analyzed (Participants) | 16
  Total active moiety after dose 3 | 25.468 (43.0)
  Total active moiety after dose 4: number analyzed (Participants) | 16
  Total active moiety after dose 4 | 23.125 (37.3)

19. Secondary Outcome: Time to Occurrence of Maximum Concentration
Description: Time to maximal observed plasma concentration (Tmax) for risperidone, 9-OH, and total active moiety after oral dosing and SC doses 1, 3 and 4.
Time Frame: Calculated over the overall dosing interval (0-12 hours on Day -1, or 0-672 hours after Dose 1, 3 or 4).
Population: PK population; actual number of participants analyzed for each period is reported
Measure: Median (Full Range); unit: hr
Arm/Group | Oral Risperidone Followed by PERSERIS
Number analyzed (Participants) | 24
hr
  Risperidone after oral dosing | 1.0 [0.50 to 4.00]
  Risperidone after Dose 1: number analyzed (Participants) | 22
  Risperidone after Dose 1 | 240.175 [4.03 to 576.23]
  Risperidone after Dose 3: number analyzed (Participants) | 16
  Risperidone after Dose 3 | 143.865 [2.03 to 503.32]
  Risperidone after Dose 4: number analyzed (Participants) | 15
  Risperidone after Dose 4 | 12.050 [2.03 to 383.87]
  9-OH after oral dosing | 1.990 [0.50 to 5.83]
  9-OH after Dose 1: number analyzed (Participants) | 22
  9-OH after Dose 1 | 204.515 [2.03 to 406.48]
  9-OH after Dose 3: number analyzed (Participants) | 16
  9-OH after Dose 3 | 182.535 [23.03 to 336.32]
  9-OH after Dose 4: number analyzed (Participants) | 15
  9-OH after Dose 4 | 118.120 [22.03 to 406.90]
  Total active moiety after oral dosing | 1.010 [0.50 to 4.00]
  Total active moiety after Dose 1: number analyzed (Participants) | 22
  Total active moiety after Dose 1 | 239.665 [4.03 to 407.87]
  Total active moiety after Dose 3: number analyzed (Participants) | 16
  Total active moiety after Dose 3 | 182.535 [23.03 to 407.03]
  Total active moiety after Dose 4: number analyzed (Participants) | 15
  Total active moiety after Dose 4 | 192.100 [6.03 to 406.90]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of informed consent through the end of study for each subject, Day 120, a total of up to 146 days including the screening and dosing stabilization periods.
Description: Adverse events (AE) were collected through a combination of systemic and non-systemic methods. AEs were collected through self-reporting by participants, and systemic methods included scheduled laboratory testing, investigator assessments of disease severity through PANSS, CGI-S and other scales, injection site assessments, ECGs, pregnancy testing for women of child-bearing potential. The one serious AE and all AEs above the frequency reporting threshold occurred in subjects receiving PERSERIS
Groups:
- Oral Risperidone Followed by PERSERIS: All participants received up to 4 monthly doses of 180 mg PERSERIS (each 180 mg dose was administered as two 90 mg SC injections). The first 3 monthly doses were administered in the abdominal region while the fourth monthly dose was administered in the back of the upper arm.
  PERSERIS: PERSERIS is an extended-release SC injectable suspension administered once-monthly
  Risperidone: Oral risperidone
  Outcome measures and adverse events were not reported by intervention, but by number of participants who experienced the adverse event. Based on narrative, it was possible to determine the timing of the serious adverse event. By nature of the adverse event, any injection site reported adverse events or outcome data occurred in participants who had received PERSERIS
Arm/Group | Oral Risperidone Followed by PERSERIS
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Risperidone Followed by PERSERIS (N=23)
increase in liver enzymes (Hepatobiliary disorders) | 1 (1) — 49 days after the last dose of PERSERIS, the participant developed increased liver enzymes reported as clinically important. The event resolved by Day 157 without intervention and was considered unrelated to study treatment by the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Risperidone Followed by PERSERIS (N=23)
upper respiratory tract infection (Infections and infestations) | 3 (3)
blood prolactin increased (Investigations) | 2 (2)
decreased appetite (Metabolism and nutrition disorders) | 2 (2)
dyskinesia (Nervous system disorders) | 2 (2)
fall (Injury, poisoning and procedural complications) | 2 (2)
headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator and Institution may have access to the Case Report Forms resulting solely from their participation in the study for purely scientific or educational purposes, but unless previously explicitly permitted in writing by the Sponsor, Principal Investigator and Institution may not use it for any publication, presentation, disclosure, or commercial purposes.

DOCUMENTS (2):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03978832/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03978832/SAP_001.pdf